CLINICAL TRIAL: NCT01218906
Title: Prospective Surveillance of Febrile Illness for Dengue-Endemic Areas in Asia
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: CYD34; U1111-1112-8378 (Other: WHO)
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Dengue Fever; Fever
Keywords: Dengue Fever Fever Dengue Infection
MeSH Terms: conditions — Dengue; Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort Population (Case ): Participants will be examined for febrile illness to diagnose dengue and to identify common causes of fever.

SUMMARY:
The purpose of this study is to detect acute febrile episodes and dengue infection in five Asian countries, to assess dengue seroprevalence, and to assess surveillance infrastructure at investigational sites in anticipation of a Phase 3 efficacy trial of a vaccine to prevent dengue infection.

The primary objectives are:

* To identify acute febrile episodes among the cohort in order to detect the presence of dengue infection.
* To develop operational infrastructure for potential Phase III dengue efficacy trial sites.
* To describe the dengue seroprevalence among the cohort at baseline and at the end of the study.

DETAILED DESCRIPTION:
All participants will make two visits to a study site, an enrollment visit and a termination visit. Additional visits will be made if febrile episodes occur: an acute visit and a convalescent visit. Participants or their parents/guardians will be contacted weekly to monitor the occurrence of febrile episodes and ensure appropriate assessment and care.

No vaccine will be provided or administered in this study.

ELIGIBILITY:
Inclusion Criteria :

* Aged 2 to 14 years on the day of inclusion and resident of the site zone
* Subject in good health, based on medical history and physical examination
* Assent form has been signed and dated by the subject (if required by local regulations), and informed consent form has been signed and dated by the parent(s) or another legally acceptable representative (and by the subject and/or an independent witness if required by local regulations)
* Subject able to attend all scheduled visits and to comply with all study procedures
* For a female of childbearing potential, use of an effective method of contraception or abstinence for at least 4 weeks prior to enrollment.

Exclusion Criteria :

* Known pregnancy at the Enrollment Visit
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding enrollment
* Planned participation in another clinical trial during the present study period
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroids therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Self-reported seropositivity for Human Immunodeficiency Virus (HIV) infection
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with study conduct or completion
* Current alcohol abuse or drug addiction that may interfere with the subject's ability to comply with study procedures
* Receipt of blood or blood-derived products in the past 3 months
* Receipt of any vaccine in the 4 weeks preceding the day of enrollment except for pandemic influenza vaccination, which may be received at least 2 weeks before enrollment
* Planned receipt of any vaccine in the 4 weeks following enrollment
* Deprived of freedom by administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Identified as employees of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members (i.e., immediate, husband, wife and their children, adopted or natural) of the employees or the Investigator.

Temporary Contraindications

A prospective subject should not be included in the study until the following condition and/or symptoms are resolved:

* Febrile illness (temperature ≥ 38.0°C) or moderate or severe acute illness/infection (according to Investigator judgment) on the day of enrollment.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants aged 2 to 14 years in 5 countries in Asia: Malaysia, Indonesia, Thailand, the Philippines and Viet Nam.
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2010-08; Primary Completion 2011-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To provide information on the incidences of febrile episodes and confirmed and probable Dengue fever, and to determine other causes of febrile episodes in the cohort population | Up to 12 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA.
Locations (11):
- Indonesia (3):
  - Bali
  - Bandung
  - Jakarta
- Malaysia (3):
  - George Town
  - Kuala Lumpur
  - Putrajaya
- Philippines (3):
  - Cebu City
  - City of Muntinlupa
  - San Pablo
- Bangkok, Thailand
- Mỹ Tho, Vietnam

REFERENCES:
- [Result] Capeding MR, Chua MN, Hadinegoro SR, Hussain II, Nallusamy R, Pitisuttithum P, Rusmil K, Thisyakorn U, Thomas SJ, Huu Tran N, Wirawan DN, Yoon IK, Bouckenooghe A, Hutagalung Y, Laot T, Wartel TA. Dengue and other common causes of acute febrile illness in Asia: an active surveillance study in children. PLoS Negl Trop Dis. 2013 Jul 25;7(7):e2331. doi: 10.1371/journal.pntd.0002331. Print 2013. PMID 23936565